CLINICAL TRIAL: NCT01191359
Title: A Multicentre Randomised Phase II Clinical Pilot Study to Compare the Pharmacodynamic Efficacy and Tolerability of the Sublingual and the Vestibular Administration Route for SLITonePLUS® Birch
Brief Title: Efficacy and Tolerability of Two Different Administration Routes With SLITonePLUS Birch
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP-B-02
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity | interventions — Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- sublingual administration (Active Comparator): oral immunotherapy with drops applied once daily by single dose containers (200 STU per dose)
  Interventions: Biological: oral immunotherapy
- vestibular administration (Active Comparator): oral immunotherapy with drops applied by single dose containers (200 STU per dose)
  Interventions: Biological: oral immunotherapy

INTERVENTIONS:
Biological: oral immunotherapy — orally applied specific immunotherapy
  Other Names: SLITone birch

SUMMARY:
Multicentre Phase II trial, comparing two different administration routes of SLITonePLUS Birch in regard to pharmacodynamic efficacy and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* A history of Birch pollen allergy
* Positive skin prick test to birch
* Positive specific IgE to birch

Exclusion criteria:

* Uncontrolled or severe asthma (FEV1<70% of predicted value in spite of adequate pharmacologic treatment)
* Previous treatment by immunotherapy with birch or a cross-reactingtree pollen allergen within the previous 5 years
* Concomitant SLIT with any allergen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic efficacy of two different administration routes of SLITonePLUS Birch | after 4, 8, 12, 24, 36 weeks of treatment
  specific antibody determination

SECONDARY OUTCOMES:
Comparison of the two administration routes with regard to safety aspects | 36 weeks
  adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bieber, MD, PhD, Principal Investigator — Universitäsklinik Bonn, Dermatology
Locations (1):
- Universitätsklinik Bonn, Dermatology, Bonn, Germany